CLINICAL TRIAL: NCT03455231
Title: Short Course Accelerated Radiation Therapy (Sharon) in Complicated Bone Metastases Palliation
Brief Title: Short Course Radiotherapy in Complicated Bone Metastases Palliation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARON-BONE
Record Dates: First submitted 2018-02-26; First posted 2018-03-06 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Palliative Care
Keywords: palliative care; complicated bone metastases; radiotherapy; pain; quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short course radiotherapy (Experimental): The radiotherapy is delivered over two days with accelerated hypo-fractionation
  Interventions: Radiation: Short course radiotherapy

INTERVENTIONS:
Radiation: Short course radiotherapy — An accelerated hypo-fractionation radiotherapy is delivered for palliation in patients with complicated bone metastases

SUMMARY:
The study wants to define the maximum tolerated dose (MTD), safety and efficacy of a short course radiation treatment in patients with complicated bone metastases.

DETAILED DESCRIPTION:
The study wants to define the maximum tolerated dose (MTD) of a conformal short course radiation treatment delivered in twice daily fractions and 2 consecutive days, and the feasibility of this fractionation in term of safety and efficacy for symptomatic palliation of complicated bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* radiologically proven complicated bone metastasis
* age > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status < 3

Exclusion Criteria:

* prior RT to the same region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  The maximum tolerated dose is defined as the dose level below the highest administered dose associated with dose limiting toxicity (DLT) in at least one third of patients

SECONDARY OUTCOMES:
Acute toxicity | 1 year
  Acute toxicity after treatment is evaluated with Common Terminology Criteria for Adverse Events (CTCAE) scale (values from 1 that represents the minimum acute toxicity to 5 that represent the maximum/severe acute toxicity).
Quality of life | 1 year
  Quality of life after treatment is evaluated according to Cancer Lineal Analog Scale (CLAS) which evaluated well-being, fatigue, and ability to perform daily activities (values range from 0 that represents the best status to 10 that represents the worst one).
Pain relief | 1 year
  Pain after the therapy is evaluated with the visual analogically scale (VAS scale). Values range from 0 (no pain) to 10 (worst possible pain).
Late toxicity | 1 year
  Late toxicity after treatment is evaluated with Toxicity criteria of the Radiation Therapy Oncology Group and the European Organization for Research and Treatment of Cancer (EORTC-RTOG scale). The values range from 1 that represents the minimum late toxicity to 5 that represent the maximum/severe late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G. Morganti, MD, Principal Investigator — Radiation Oncology Center, Department of Experimental, Diagnostic and Specialty Medicine - DIMES, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Capuccini J, Macchia G, Farina E, Buwenge M, Genovesi D, Caravatta L, Nguyen NP, Cammelli S, Cilla S, Wondemagegnhu T, Uddin AFMK, Aziz Sumon M, Cellini F, Valentini V, Deodato F, Morganti AG. Short-course regimen of palliative radiotherapy in complicated bone metastases: a phase i-ii study (SHARON Project). Clin Exp Metastasis. 2018 Oct;35(7):605-611. doi: 10.1007/s10585-018-9931-9. Epub 2018 Aug 18. PMID 30121938